CLINICAL TRIAL: NCT00003950
Title: A Phase II Trial of Irinotecan (CPT-11) and Cyclosporine in Patients With 5-FU Refractory Advanced Colorectal Cancer
Brief Title: Irinotecan and Cyclosporine in Treating Patients With Metastatic, Advanced or Locally Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9824; UCCRC-T98-0049; NCI-T98-0049
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cyclosporine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPT-11 with Cyclosporine (Experimental): Each cycle lasts 6 weeks. Administration of cyclosporine and CPT-11 weekly for 4 weeks followed by a 2 week 'rest' period with no drug given. Cyclosporine is given by IV infusion at a dose of 5 mg/kg. CPT-11 is given by IV infusion at a dose of 60 mg/m2.
  Interventions: Drug: cyclosporine; Drug: CPT-11

INTERVENTIONS:
Drug: cyclosporine
  Other Names: Sandimmune®, Restatis®
Drug: CPT-11
  Other Names: Irinotecan, Camptosar®

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Cyclosporine may relieve the diarrhea caused by irinotecan.

PURPOSE: Phase II trial to study the effectiveness of irinotecan and cyclosporine in treating patients who have metastatic, advanced, or locally recurrent colorectal cancer that has not responded to fluorouracil.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with metastatic, advanced, or locally recurrent fluorouracil refractory adenocarcinoma of the colon or rectum treated with irinotecan and cyclosporine. II. Determine antitumor activity, safety, tolerance, and toxicity of this combination treatment in these patients.

OUTLINE: This is a multicenter study. Patients receive cyclosporine IV over 6 hours and irinotecan IV over 90 minutes weekly for 4 weeks. Courses repeat every 6 weeks. Patients receive at least 2 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 15-45 patients will be accrued for this study over 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic, advanced, or locally recurrent fluorouracil (5-FU) refractory adenocarcinoma of the colon or rectum Progression of disease within 6 months of receiving adjuvant 5-FU based chemotherapy OR Progression of disease during or following completion of 5-FU based chemotherapy for metastatic disease No more than 1 failure with a 5-FU regimen for recurrent, advanced, or metastatic disease Failure on 5-FU adjuvant therapy must accompany failure on 5-FU therapy for metastatic disease Bidimensionally measurable disease CNS metastases allowed only with measurable disease in other sites Prior treatment for CNS metastases required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3500/mm3 Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST and ALT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: No other significant, uncontrolled underlying medical or psychiatric condition No serious active infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Neurologically stable No other prior malignancy within past 5 years except curatively treated nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics Prior adjuvant fluorouracil (5-FU) allowed No more than 2 prior 5-FU regimens (no more than 1 for recurrent or metastatic disease) No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy (except contraceptives or replacement steroids) No concurrent IV steroids Radiotherapy: Prior radiotherapy allowed if measurable disease outside radiation port At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: No concurrent anticonvulsant therapy No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2000-01; Primary Completion 2001-12 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Reduction in occurrences of severe diarrhea due to CPT-11 administration | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana

REFERENCES:
- [Result] Desai AA, Kindler HL, Taber D, Agamah E, Mani S, Wade-Oliver K, Ratain MJ, Vokes EE. Modulation of irinotecan with cyclosporine: a phase II trial in advanced colorectal cancer. Cancer Chemother Pharmacol. 2005 Oct;56(4):421-6. doi: 10.1007/s00280-005-1020-5. Epub 2005 May 13. PMID 15895230